CLINICAL TRIAL: NCT07185009
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-Controlled, Phase 3 Maintenance Study to Evaluate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Maintenance Study to Investigate the Efficacy and Safety of Duvakitug in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: SUNSCAPE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18359; 2025-521038-27 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Duvakitug - dose 1 (Experimental): Subcutaneous (SC) injection as per protocol
  Interventions: Drug: Duvakitug
- Duvakitug - dose 2 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Duvakitug - dose 3 (Experimental): SC injection as per protocol
  Interventions: Drug: Duvakitug
- Placebo (Placebo Comparator): SC injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duvakitug — Pharmaceutical form: Injection solution Route of administration: SC injection
  Arms: Duvakitug - dose 1; Duvakitug - dose 2; Duvakitug - dose 3
Drug: Placebo — Pharmaceutical form:Injection solution-Route of administration:SC injection
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 3 maintenance study to evaluate the efficacy and safety of duvakitug in participants with moderately to severely active Ulcerative Colitis (UC).

Study details include:

The study duration may be up to 286 weeks including:

* 40-week Pivotal Maintenance Sub-Study
* 240-week Open-Label Extension (OLE) Sub-Study
* 45-day Follow-up Visit Note: For the participants who do not enroll into OLE Sub-Study, the duration will be up to 46 weeks, including the 40-week maintenance period and a 45-day follow-up visit.

The treatment duration may be up to 280 weeks including:

* 40 weeks in Pivotal Maintenance Sub-Study
* 240 weeks in OLE Sub-Study

The total number of on-site visit will be up to 32:

* 21 visits in the Pivotal Maintenance Sub-Study.
* 11 visits in the OLE Sub-Study.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥18 and ≤80 years of age at Baseline. (Where locally permissible, participants 16 to <18 years of age who meet the definition of Tanner stage 5 for development)
* Pivotal Maintenance Sub-Study: Participants who achieved clinical response and completed endoscopy at the end of SUNSCAPE-1
* OLE Sub-Study: Participants who complete the Pivotal Maintenance Sub-Study or participation in the TV48574-IMM-20038 Study

Exclusion Criteria:

* Participants with medical or compliance conditions that are deemed unsuitable for the study by the investigator
* Participants with a known hypersensitivity to duvakitug that makes the participant unsuitable for the study by the investigator

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 671 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2028-09-21 (Estimated); Study Completion 2033-04-28 (Estimated)

PRIMARY OUTCOMES:
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving clinical remission by modified Mayo Score (mMS). | Week 40
  Mayo Score is a composite index designed to measure UC disease activity. The score ranges from 0 to 9 with higher scores indicating greater disease severity. Clinical remission is defined as mMS score of 0 to 2, including SFS of 0 or 1, RBS of 0, and mMES of 0 or 1 (score of 1 modified to exclude friability)

SECONDARY OUTCOMES:
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with endoscopic improvement. | Week 40
  Endoscopic improvement is defined as mMES of 0 or 1 (score of 1 excludes friability).
  Endoscopies were assessed by a blinded central reader and scored according to the following scale: 0 = Normal or inactive disease; 1 = Mild disease (erythema, decreased vascular pattern); 2 = Moderate disease (marked erythema, lack of vascular pattern, any friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration).
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving histologic endoscopic mucosal improvement. | Week 40
  Histological endoscopic mucosal improvement is defined as MES of 0 or 1 without the evidence of friability and Geboes Score ≤3.1.
  The Geboes score has 6 grades: Grade 0, structural change only; Grade 1, chronic inflammation; Grade 2, lamina propria neutrophils and eosinophils; Grade 3, neutrophils in epithelium; Grade 4, crypt destruction; and Grade 5, erosions or ulceration.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with corticosteroid-free clinical remission. | Week 40
Proportion of participants with no bowel urgency. | Week 40
  The NRS for bowel urgency is a patient-reported tool designed to measure the severity of bowel urgency-the sudden or immediate need to have a bowel movement-experienced in the past 24 hours. This tool utilizes an 11-point scale for evaluation, where 0 represents "no urgency" and 10 signifies the "worst possible urgency".
Pivotal Maintenance Sub-Study Cohort 1: Change from Baseline in PROMIS-Fatigue Short Form 7a T-score. | Baseline, Week 40
  The PROMIS Fatigue Short Form 7a uses a 5-point Likert scale for each of its 7 items, resulting in a raw score range of 7 to 35. This raw score is then converted into a T-score, with a mean of 50 and a standard deviation of 10, based on US national norms. Higher Tscores indicate greater fatigue.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with endoscopic remission. | Week 40
  Endoscopic remission is defined as mMES of 0.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving clinical remission by mMS, in the subset of participants who achieved clinical remission by mMs at the end of induction period (maintenance of clinical remission). | Week 40
  Clinical response is defined as a decrease from baseline in the mMS of ≥2 points and at least a 30% reduction from baseline, and a decrease in RB subscore of ≥1 or an absolute RB subscore of 0 or 1.
  Mayo Score is a composite index designed to measure UC disease activity. The score ranges from 0 to 9 with higher scores indicating greater disease severity.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with no abdominal pain by Numerical Rating Scale (NRS). | Week 40
  The abdominal pain NRS is a tool to rate the severity of abdominal pain over the past 24 hours using a score of 0 ("no pain") to 10 ("worst possible pain").
Pivotal Maintenance Sub-Study Cohort 1: Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score | Week 40
  IBDQ is a tool to the quality of life of individuals suffering from IBD. The total score ranges from 32 to 224, with higher scores correlating to a better quality of life.
Pivotal Maintenance Sub-Study Cohort 1: Incidence of UC-related hospitalizations. | Week 0 through Week 40
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants with symptomatic (stool-frequency sub score [SFS] and = rectal bleeding sub score [RBS]) remission. | Week 40
  Symptomatic response is defined as ≥30% decrease from baseline in the composite clinical endpoint of the sum of SFS and RBS.
Pivotal Maintenance Sub-Study Cohort 1: Proportion of participants achieving clinical remission and no steroid use from the baseline to the time of endpoint analysis. | Week 40
Pivotal Maintenance Sub-Study Cohort 1: Incidence of Treatment-Emergent Adverse Events (TEAEs), TEAEs of Special Interest, Treatment-Emergent Serious Adverse Events (TESAEs), and TEAEs leading to permanent study intervention discontinuation. | Week 0 through 45 days after last dose
Pivotal Maintenance Sub-Study Cohort 1: Serum concentration of duvakitug measured over time. | Week 0 through Week 40
Pivotal Maintenance Sub-Study Cohort 1: Incidence of treatment-emergent Anti-Drug Antibodies (ADA) against duvakitug. | Week 0 through Week 40
Open-Label Extension Sub-Study: Incidence of Treatment-Emergent Adverse Events (TEAEs), TEAEs of Special Interest, Treatment-Emergent Serious Adverse Events (TESAEs), and TEAEs leading to permanent study intervention discontinuation. | Week 40 of pivotal maintenance through 45 days after last dose

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Royal Palm Clinical Research - Site Number: 8400065, Fort Myers, Florida
  - Clinical Research of Osceola - Site Number: 8400013, Kissimmee, Florida
  - Delta Research Partners - Site Number: 8400087, Monroe, Louisiana
  - BVL Clinical Research - Site Number: 8400005, Liberty, Missouri

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org